CLINICAL TRIAL: NCT05595187
Title: Concomitant Tricuspid Repair in Patients With Left Heart Surgery: Randomized Controlled Trial
Brief Title: Concomitant Tricuspid Repair in Patients With Left Heart Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of Cardiovascular Surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JPH-2022
Record Dates: First submitted 2022-10-23; First posted 2022-10-26 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Tricuspid Regurgitation; Mitral Regurgitation; Cardiopulmonary Bypass
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Mitral Valve Insufficiency

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tricuspid repair (Experimental): Tricuspid repair techniques included suture placement and the type of prosthetic annuloplasty with specified the use of an approved rigid, incomplete, nonplanar, and undersized (ranging 26, 28, or 30, 32, 34 mm) ring.
  Interventions: Device: Tricuspid repair
- Blank control (No Intervention)

INTERVENTIONS:
Device: Tricuspid repair — Tricuspid repair included suture placement and the type of prosthetic annuloplasty.
  Arms: Tricuspid repair

SUMMARY:
Tricuspid regurgitation is common in patients with severe left heart diseases, such as degenerative mitral regurgitation. However, the evidence base is insufficient to inform a decision about whether to perform concomitant tricuspid-valve repair during left heart surgery in patients who have mild tricuspid regurgitation. To inform decision making, we will conduct a multicenter, randomized trial to assess the benefits and risks of tricuspid-valve repair at the time of left heart diseases in patients with mild tricuspid regurgitation who were undergoing surgery for left heart surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing left heart valve surgery with mild tricuspid regurgitation;
2. Patients aged 18-80 years;
3. Agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Infective endocarditis within 3 months;
2. Primary tricuspid regurgitation;
3. Isolated tricuspid regurgitation
4. Lactating women and suspected pregnant or pregnant women;
5. Patients with mental disorders, drug and alcohol dependence;
6. Those who participated in other clinical trials one month before the trial;
7. Refusal to participate in this study without informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite of adverse cardiovascular events | 2 years after surgery at follow-up
  a composite of reoperation for tricuspid regurgitation, progression of tricuspid regurgitation from baseline by two grades or the presence of severe tricuspid regurgitation, or death.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: Undecided